CLINICAL TRIAL: NCT00819104
Title: A Five-arm, Randomised, Open Label, Multi-centre, Prospective Study to Compare the Efficacy, Safety and Tolerability of Metoprolol XL Plus Amlodipine Combination (Selomax TM) With Metoprolol XL and Amlodipine as Individual Components in Management of Hypertension in Indian Patients.
Brief Title: A Study to Compare the Efficacy, Safety and Tolerability of Selomax With Its Individual Components
Acronym: MARS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Dr. Paurus M Irani; VP Medical & Regulatory, AstraZeneca Pharmaceuticals India Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4022L00006
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Primary Hypertension
Keywords: Primary hypertension; Metoprolol XL; Amlodipine
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): FDC of Metoprolol XL 50mg + Amlodipine 5mg
  Interventions: Drug: Metoprolol XL 50mg + Amlodipine 5mg
- 2 (Experimental): FDC of Metoprolol XL 25mg + Amlodipine 2.5mg
  Interventions: Drug: Metoprolol XL 25 mg + Amlodipine 2.5mg
- 3 (Active Comparator): Extended release Metoprolol succinate
  Interventions: Drug: Metoprolol XL 50mg
- 4 (Active Comparator): Extended release Metoprolol succinate
  Interventions: Drug: Metoprolol XL 25 mg
- 5 (Active Comparator): Amlodipine 5mg in immediate release formulation
  Interventions: Drug: Amlodipine 5mg

INTERVENTIONS:
Drug: Metoprolol XL 50mg + Amlodipine 5mg — tablet,oral,OD,8 weeks
  Other Names: Selomax 50/5
  Arms: 1
Drug: Metoprolol XL 25 mg + Amlodipine 2.5mg — tablet,oral,OD,8 weeks
  Other Names: Selomax 25/2.5
  Arms: 2
Drug: Metoprolol XL 50mg — tablet,oral,OD,8 weeks
  Other Names: Revelol XL
  Arms: 3
Drug: Metoprolol XL 25 mg — tablet,oral,OD,8 weeks
  Other Names: Revelol XL
  Arms: 4
Drug: Amlodipine 5mg — tablet,oral,OD,8 weeks
  Other Names: Amlogard
  Arms: 5

SUMMARY:
This is a randomised, open-label; parallel group, multicentric study comparing the efficacy and safety of fixed-dose-combinations of Metoprolol XL plus Amlodipine with individual components of the combination. SelomaxTM50/5 will also be compared with SelomaxTM 25/2.5 in lowering of BP (SBP and DBP) in Indian patients with essential hypertension.Male and female patients of essential hypertension aged between 18-80 years will be studied. The patients should not have a history of prior cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of hypertension (primary) , as judged by 2 BP measurements before randomisation
* Those who have given their written consent for the study.

Exclusion Criteria:

* Patients of other forms of hypertension (other than primary)
* Those who have consistently BP > /=180/120mmHg
* Patients with a prior history of chest pain, heart attacks, conduction defects and strokes.
* Patients of diabetes requiring insulin,asthma and kidney diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2008-11; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in BP with Selomax™ 50/5 at the end of the randomisation treatment period. | 8 weeks

SECONDARY OUTCOMES:
Change in BP (SBP,DBP & mean BP) with SelomaxTM 25/2.5 at the end of the randomisation period. | 8 weeks
Change in the heart rate,Number of responders & control rates. | 8 weeks
Incidence of adverse events (serious and non-serious) in each arm.Change in hemogram, serum chemistry (Liver function tests (LFT), Renal function tests (RFT), plasma lipids, Blood Glucose, HbA1c), and Ur.albumin | 8 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- India (11):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Calicut, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Delhi, National Capital Territory of Delhi
  - Research Site, Jaipur, Rajasthan
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
  - Research Site, Bangalore